CLINICAL TRIAL: NCT06529458
Title: Effects of Acupressure and Aromatherapy Applied to Patients Receiving Chemotherapy on Severity of Nausea and Vomiting, Anxiety and Comfort Levels
Brief Title: Effects of Acupressure and Aromatherapy on Nausea and Vomiting Severity, Anxiety and Comfort Level
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Setenay Batır (Other Government)
Responsible Party: Sponsor-Investigator, Setenay Batır, Lecturer, Kayseri City Hospital
Organization: Kayseri City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Acupress and aromatherapy
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer Patients Receiving Chemotherapy
Keywords: Chemotherapy; Acupressure; Aromatherapy; Nausea Vomiting Severity; Anxiety; Comfort Level
MeSH Terms: conditions — Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention 1 Group (Experimental): The researcher will apply pressure to the P6 acupressure point on both wrists for approximately 5 minutes at the same time as chemotherapy. He will also have the patient or a relative repeat the method and do it at home three times a day before meals for 5 days.
  Interventions: Other: Intervention 1 Group
- Intervention 2 Group (Experimental): The researcher will apply drops of ginger oil to the P6 acupressure point on both wrists for approximately 5 minutes at the same time as chemotherapy, using circular motions. At the same time, the researcher will have the patient or a relative repeat the method and apply it at home three times a day before meals for 5 days.
  Interventions: Other: Intervention 2 Group
- Control Group (Other): No interference will be made
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Intervention 1 Group — The researcher will apply pressure to the P6 acupressure point on both wrists for approximately 5 minutes at the same time as chemotherapy. He will also have the patient or a relative repeat the method and do it at home three times a day before meals for 5 days.
  Arms: Intervention 1 Group
Other: Intervention 2 Group — The researcher will apply drops of ginger oil to the P6 acupressure point on both wrists for approximately 5 minutes at the same time as chemotherapy, using circular motions. At the same time, the researcher will have the patient or a relative repeat the method and apply it at home three times a day before meals for 5 days.
  Arms: Intervention 2 Group
Other: Control Group — No interference will be made
  Arms: Control Group

SUMMARY:
The aim of the researchers is to evaluate the effects of acupressure applied to the p6 region for 5 days and acupressure applied by applying ginger oil on the severity of nausea and vomiting, anxiety and comfort levels in patients receiving chemotherapy. The study is a randomized, controlled experimental study.

It will be conducted on patients diagnosed with breast cancer who are receiving treatment at the Erciyes University Health Application and Research Center Nazende-Nuri Özkaya Oncology Day Treatment Center. A total of 60 patients, 20 patients in control, 20 patients in Intervention 1 and 20 patients in Intervention 2 who meet the inclusion criteria, will be included in the sample according to the block randomization list created in the computer environment. Attention will be paid to ensure that the patients have similar characteristics such as being diagnosed with breast cancer, receiving chemotherapy for the first time, using the same chemotherapy drugs and the same antiemetic drugs (Adriablastin, Cyclophosphamide, Kytril), gender and age. No application will be made to the control group.

Data; Data will be collected using the Informed Consent Form, Patient Introduction Form, Visual Analog Scale (VAS), Rhodes Nausea, Vomiting and Retching Index (INVR), General Comfort Scale-Short Form, State-Trait Anxiety Inventory (STAI), Patient Monitoring Schedule-Researcher Form, Acupressure Application Protocol, Acupressure and Aromatherapy Application Protocol.

DETAILED DESCRIPTION:
Cancer is a major public health problem that threatens life and health. The aim of cancer treatment is to extend the life span of the individual and improve the quality of life. The process of cancer treatment is long and difficult. Cancer patients face various physical (hair loss, nausea, vomiting, pain, fatigue, loss of appetite, malnutrition and weakness) and psychological complications (depression, stress and anxiety) that reduce their quality of life during the treatment process. Despite the use of various treatments such as surgery, chemotherapy, hormone therapy, radiotherapy, immunotherapy and biological therapy in cancer treatment today, patients still complain of many physical and psychological complications. Nausea and vomiting, which are among the side effects of treatment, are the most common and disturbing symptoms. Despite the development of drug treatments in recent years, nausea and vomiting due to chemotherapy is seen in an average of 38%-80% of patients. Nausea due to cancer treatments can be acute (occurring within 24 hours of treatment), delayed (occurring after the first 24 hours of treatment and continuing for 1-4 days), anticipatory (occurring due to conditioning before or during treatment), breakthrough nausea and/or vomiting (occurring despite prophylactic medications and requiring additional treatment), refractory (unresponsive/persistent to treatment), and chronic vomiting. Nausea and vomiting are known to cause serious problems such as fluid and electrolyte imbalance, weight loss, dehydration, and malnutrition, as well as negatively impacting patients' daily activities and quality of life. Uncontrolled nausea and vomiting can also cause patients to delay or refuse treatment. Anxiety, which occurs during the long and difficult treatment process of cancer, is often difficult to define and treat. Some events that may cause anxiety in cancer patients include hearing the diagnosis, receiving chemotherapy, undergoing surgery, receiving radiation therapy, and discussing family problems. Anxiety symptoms have been reported to be observed in 20% to 60% of cancer patients. Today, traditional complementary and alternative medicine treatments are widely used to relieve cancer symptoms due to their organic nature, fewer complications, and lower costs. Acupressure is a treatment method that has been used in Traditional Chinese Medicine for 5000 years. In the literature, acupressure applications have been used to improve sleep quality, relieve pain related to childbirth and cancer, reduce fatigue, depression, and anxiety, and relieve nausea and vomiting. Acupressure can be applied to the P6 acupuncture point with pressure methods using a wrist band or fingers. The wrist band comes in different sizes and has been developed with a round hemisphere on its inner surface that can apply pressure to the P6 point. Although the effect of acupressure on nausea and vomiting has not been fully explained, it is thought that it reduces nausea and vomiting by increasing the release of neurohormones and neurotransmitters (beta endorphin, serotonin, histamine) and regulating blood circulation as a result of stimulating acupressure points. Another study has indicated that acupressure increases the energy flow on the meridians and thus reduces nausea and vomiting. In the studies conducted by Genç and Tan with breast cancer patients, it was reported that pressure applied to the P6 point with acupressure technique was effective in reducing nausea. Another study conducted on breast cancer patients indicated that acupressure application to the P6 point caused a decrease in nausea, vomiting and anxiety levels of the patients and emphasized that more studies should be conducted on this subject. In another study, patients were divided into two groups for acupressure application: pressure (n = 22) and wrist band (n = 22). Acupressure was applied to both wrists for two minutes using the finger pressure method and for fifteen minutes using a wrist band. The number and severity of nausea and vomiting were found to be statistically significantly lower in the pressure and wrist band groups compared to placebo applications. It was found that additional antiemetic drug use was statistically significantly higher in the placebo groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years of age or older,
* Understand and communicate in Turkish,
* Those who are diagnosed with breast cancer and receive their first course of chemotherapy,
* Those who are receiving platinum group chemotherapeutic agents (Adriablastin, Cyclophosphamide) that have a high emotogenic effect,
* Those who are not pregnant and not planning to be pregnant,
* Those whose disease stage is at most stage III,
* Those who do not have any psychiatric disorders,
* Those who do not have wounds, lesions, etc. in the areas where acupressure will be applied

Exclusion Criteria:

* Individuals who have another disease that may affect nausea and vomiting,
* Those who are allergic to ginger or are bothered by its smell,
* Those who receive simultaneous radiotherapy,
* Those who use other complementary and integrated treatment practices during the treatment process will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-29 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Day 1
  The scale consists of a horizontal line 100 mm/10 cm long. At the left end of the line is 0 "No nausea", while at the right end is 10 "Severe nausea". The patient will be asked to mark the point on the line that will accurately reflect their nausea. In patient selection, 5 mm and below on the scale will be evaluated as "no nausea" and all values above will be evaluated as "experiencing nausea".
Rhodes Index of Nausea, Vomiting ve Retching- INVR | Day 1
  This index measures the number of nausea, vomiting and retching episodes and the distress experienced by individuals in the last 12 hours using a Likert-type assessment. The index consists of 8 questions. Each answer is scored as "0" for the least distress; "4" for the most distress.
General Comfort Scale-Short Form | Day 1
  The scale consists of three sub-dimensions: relief (1-9 items), relaxation (10-18 items) and superiority (19-28 items). The lowest score that can be obtained from the scale is 28 and the highest score is 168. As the score obtained from the scale decreases, it indicates that the individual's comfort level is low. The lowest value "1" indicates low comfort and "6" indicates high comfort level.
State-Trait Anxiety Inventory | Day 1
  While the state anxiety scale only provides information about what is felt at that moment, the trait anxiety scale was developed to measure what has been felt over the last 7 days. In interpreting the scores, the total score obtained from both scales varies between 20 and 80. A high score indicates a high level of anxiety, and a low score indicates a low level of anxiety.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | Immediately after chemotherapy treatment
  The scale consists of a horizontal line 100 mm/10 cm long. At the left end of the line is 0 "No nausea", while at the right end is 10 "Severe nausea". The patient will be asked to mark the point on the line that will accurately reflect their nausea. In patient selection, 5 mm and below on the scale will be evaluated as "no nausea" and all values above will be evaluated as "experiencing nausea".

OTHER OUTCOMES:
Visual Analog Scale (VAS) | One day after chemotherapy treatment
  The scale consists of a horizontal line 100 mm/10 cm long. At the left end of the line is 0 "No nausea", while at the right end is 10 "Severe nausea". The patient will be asked to mark the point on the line that will accurately reflect their nausea. In patient selection, 5 mm and below on the scale will be evaluated as "no nausea" and all values above will be evaluated as "experiencing nausea".
Rhodes Index of Nausea, Vomiting ve Retching- INVR | One day after chemotherapy treatment
  This index measures the number of nausea, vomiting and retching episodes and the distress experienced by individuals in the last 12 hours using a Likert-type assessment. The index consists of 8 questions. Each answer is scored as "0" for the least distress; "4" for the most distress.
Visual Analog Scale (VAS) | 2nd, 3rd, 4th day after chemotherapy treatment
  The scale consists of a horizontal line 100 mm/10 cm long. At the left end of the line is 0 "No nausea", while at the right end is 10 "Severe nausea". The patient will be asked to mark the point on the line that will accurately reflect their nausea. In patient selection, 5 mm and below on the scale will be evaluated as "no nausea" and all values above will be evaluated as "experiencing nausea".
Visual Analog Scale (VAS) | 5th day after chemotherapy treatment
  The scale consists of a horizontal line 100 mm/10 cm long. At the left end of the line is 0 "No nausea", while at the right end is 10 "Severe nausea". The patient will be asked to mark the point on the line that will accurately reflect their nausea. In patient selection, 5 mm and below on the scale will be evaluated as "no nausea" and all values above will be evaluated as "experiencing nausea".
General Comfort Scale-Short Form | 5th day after chemotherapy treatment
  The scale consists of three sub-dimensions: relief (1-9 items), relaxation (10-18 items) and superiority (19-28 items). The lowest score that can be obtained from the scale is 28 and the highest score is 168. As the score obtained from the scale decreases, it indicates that the individual's comfort level is low. The lowest value "1" indicates low comfort and "6" indicates high comfort level.
State-Trait Anxiety Inventory | 5th day after chemotherapy treatment
  While the state anxiety scale only provides information about what is felt at that moment, the trait anxiety scale was developed to measure what has been felt over the last 7 days. In interpreting the scores, the total score obtained from both scales varies between 20 and 80. A high score indicates a high level of anxiety, and a low score indicates a low level of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Setenay Batır, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Genc F, Tan M. The effect of acupressure application on chemotherapy-induced nausea, vomiting, and anxiety in patients with breast cancer. Palliat Support Care. 2015 Apr;13(2):275-84. doi: 10.1017/S1478951514000248. Epub 2014 Apr 30. PMID 24787745